CLINICAL TRIAL: NCT03409900
Title: Lumbar Plexus Block Versus Quadratus Lumborum Block for Primary Anterior Total Hip Arthroplasty: A Non-inferiority Trial
Brief Title: Lumbar Plexus Block Versus Quadratus Lumborum Block for Primary Anterior Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00048845
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Total Hip Arthroplasty
Keywords: Lumbar Plexus Block; Quadratus Lumborum Block; Direct Anterior Approach; Post-Operative; Pain Management
MeSH Terms: conditions — Osteoarthritis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPB Unilateral DAA THA (Experimental): Patients will be randomized to receive either a LPB or QLB for post-operative analgesia. Randomization to either LPB or QLB will occur via block randomization using sealed sequentially numbered opaque envelopes that will correspond to the order with which patients are enrolled. Patients and research assistants will be blinded to their randomization by administration of intravenous sedation (titrated to patient comfort), utilization of ultrasonography to visualize pertinent structures for both blocks, and by the nature of the block technique themselves both being in close proximity on the posterior lower back.
  Interventions: Other: LPB
- QLB Unilateral DAA THA (Experimental): Patients will be randomized to receive either a LPB or QLB for post-operative analgesia. Randomization to either LPB or QLB will occur via block randomization using sealed sequentially numbered opaque envelopes that will correspond to the order with which patients are enrolled. Patients and research assistants will be blinded to their randomization by administration of intravenous sedation (titrated to patient comfort), utilization of ultrasonography to visualize pertinent structures for both blocks, and by the nature of the block technique themselves both being in close proximity on the posterior lower back.
  Interventions: Other: QLB

INTERVENTIONS:
Other: LPB — The LPB will be performed in a lateral position, but modified to utilize ultrasound guidance to enhance our ability to quickly and safely locate the lumbar plexus as well as to avoid unblinding with regard to the traditional landmark LPB technique. For both LPB and QLB a TOTAL DOSE of 20 cc of the following local anesthetic mixture will be administered: Ropivacaine 0.2% and Epinephrine - 2.5 mcg/cc (1:400,000 concentration).
  Other Names: Lumbar Plexus Block
  Arms: LPB Unilateral DAA THA
Other: QLB — The QLB will be performed in a lateral position in a manner consistent with the technique first described by Børglum. For both LPB and QLB a TOTAL DOSE of 20 cc of the following local anesthetic mixture will be administered: Ropivacaine 0.2% and Epinephrine - 2.5 mcg/cc (1:400,000 concentration).
  Other Names: Quadratus Lumborum Block
  Arms: QLB Unilateral DAA THA

SUMMARY:
Total hip arthroplasty (THA) is one of the most successful orthopedic procedures to effectively relieve pain and restore function in patients with end stage osteoarthritis. In an attempt to accelerate recovery many orthopedic surgeons have opted to utilize a direct anterior approach (DAA) as opposed to the more traditional posterolateral approach (PLA). The literature supports that DAA is superior to PLA with regard to lower blood loss, less pain, shorter hospital stay, and faster rehabilitation. Traditionally the study team has performed Lumbar Plexus blocks (LPB) to provide post-operative analgesia for total hip arthroplasty. The quadratus lumborum block (QLB) is a newer regional analgesic technique that may be as effective as LPB at providing pain control following DAA hip arthroplasty. This study is designed to compare the efficacy, with regards to post-operative pain management, between LPB and QLB following a DAA total hip arthroplasty.

DETAILED DESCRIPTION:
In an attempt to accelerate recovery many orthopedic surgeons have opted to utilize a direct anterior approach (DAA) as opposed to the more traditional posterolateral approach (PLA) in regards to total hip arthroplasty (THA). The DAA technique involves dissection of muscular planes for insertion of components resulting in less tissue damage as compared to PLA. Traditionally the study team has performed Lumbar Plexus blocks (LPB) to provide post-operative analgesia for total hip arthroplasty. This technique works well for the traditionally performed PLA in that the hip joint and incision site are within the analgesic distribution of the LPB. Conversely, the DAA utilizes an anterior incision that overlies the L1 and L2 dermatomes as opposed to the lower lumbar dermatomes of the PLA incision. When performing LPB it has been the study team's clinical experience that it is rare to achieve analgesia in the proximal distribution of the lumbar plexus resulting in apparent sparing of the L1 and L2 nerve root distributions. The quadratus lumborum block (QLB) is a newer regional analgesic technique that may be as effective as LPB at providing pain control following DAA hip arthroplasty. The QLB is thought to provide analgesia by blocking both the lateral and anterior cutaneous branches of T7 through L4. This degree of dermatomal coverage suggests that QLB could be an efficacious alternative to LPB for DAA hip arthroplasty. It is hypothesized that the QLB will provide equivalent analgesia when compared to the LPB as determined by a comparison of verbal reported pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the ages of 18 and 95 years undergoing a primary elective, unilateral DAA total hip arthroplasty.

Exclusion Criteria:

* If the patient uses more than 40mg of Oxycodone equivalents per 24 hours or is on extended release opioid formulations.
* Indication for surgery is secondary to trauma and/or hip fracture
* If there is a contraindication to the performance of a regional block
* Concomitant anticoagulation use or documented coagulopathy
* Infectious or dermatologic conditions in the area of block placement that would otherwise increase the risk of peripheral nerve blockade
* Presence of progressive neurologic deficit effecting peripheral nerves
* Allergy or adverse reaction to study drugs to include: fentanyl, epinephrine, and amide local anesthetics
* American Society of Anesthesia Physical Classification score > or = to 4
* Allergies to study drugs other than local anesthetic
* BMI > 40
* Patient refusal
* Pregnancy
* Institutionalized individuals
* Extremes of age: Age > 95 or < 18
* Non English speaking or inability to reliably participate in the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Verbal numeric pain score with hip flexion at 6hrs (Numeric Rating Scale (NRS)) | 6 hours post block
  Quantified on an 10 point pain scale with 0 representing "no pain" and 10 representing "worst pain imaginable". Higher scores denotes worse outcomes.

SECONDARY OUTCOMES:
Time to first analgesic | During hospitalization, up to 24hrs
  Time from PACU discharge to first requested analgesic
Total opioid consumption over 24 hours | 24 hrs post block
  Total opioid consumption in the first 24hrs
Verbal numeric pain score at 6hrs at rest (NRS) | 6hrs post block
  Quantified on an 10 point pain scale with 0 representing "no pain" and 10 representing "worst pain imaginable". Higher scores denotes worse outcomes.
Verbal numeric pain score at rest and with movement at 24hrs post block | 24hrs post block
  Quantified on an 10 point pain scale with 0 representing "no pain" and 10 representing "worst pain imaginable". Higher scores denotes worse outcomes.
Ability to straight leg raise on POD1 | Post operative day 1
  Is the patient able to perform an unassisted straight leg raise
Rates of opioid related side effects (nausea, vomiting, pruritis) | Within 24hrs post block
  Has the patient had any nausea, vomiting, or pruritis within the first 24hrs
Patient satisfaction utilizing a Likert-scale questionnaire | Post operative day 1
  A patient satisfaction survey to administered on post operative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Edwards, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-12-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03409900/ICF_000.pdf